CLINICAL TRIAL: NCT01031901
Title: Topical Rapamycin Therapy to Alleviate Cutaneous Manifestations of Tuberous Sclerosis Complex and Neurofibromatosis 1
Brief Title: Topical Rapamycin Therapy to Alleviate Cutaneous Manifestations of Tuberous Sclerosis Complex (TSC) and Neurofibromatosis I (NF1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Principal Investigator, Mary Kay Koenig, Assistant Professor, Pediatrics-Neurology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-09-0259
Record Dates: First submitted 2009-12-10; First posted 2009-12-15 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Tuberous Sclerosis; Neurofibromatoses; Angiofibroma; Neurofibroma
Keywords: Tuberous Sclerosis; Neurofibromatoses; Angiofibroma; Neurofibroma; Sirolimus
MeSH Terms: conditions — Tuberous Sclerosis; Neurofibromatoses; Angiofibroma; Neurofibroma | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- TSC Placebo Arm (Placebo Comparator): TSC subjects will apply a study product containing polyvinylidene fluoride coating alone to facial angiofibromas
  Interventions: Drug: Skincerity
- TSC 1% Arm (Experimental): TSC subjects will apply a study product containing polyvinylidene fluoride coating plus 1 mg of sirolimus/rapamycin to facial angiofibromas
  Interventions: Drug: Skincerity plus sirolimus/rapamycin
- TSC 5% Arm (Experimental): TSC subjects will apply a study product containing polyvinylidene fluoride coating plus 5 mg of sirolimus/rapamycin to facial angiofibromas
  Interventions: Drug: Skinercity plus sirolimus/rapamycin
- NF1 Placebo Arm (Placebo Comparator): NF1 subjects will apply a study product containing polyvinylidene fluoride coating alone to cutaneous neurofibromas
  Interventions: Drug: Skincerity
- NF1 1% Arm (Experimental): NF1 subjects will apply a study product containing polyvinylidene fluoride coating plus 1 mg of sirolimus/rapamycin to cutaneous neurofibromas
  Interventions: Drug: Skincerity plus sirolimus/rapamycin
- NF1 5% Arm (Experimental): NF1 subjects will apply a study product containing polyvinylidene fluoride coating plus 5 mg of sirolimus/rapamycin to cutaneous neurofibromas
  Interventions: Drug: Skinercity plus sirolimus/rapamycin

INTERVENTIONS:
Drug: Skincerity — Study subjects will apply a study product containing polyvinylidene fluoride coating alone to either facial angiofibromas or cutaneous neurofibromas
  Arms: NF1 Placebo Arm; TSC Placebo Arm
Drug: Skincerity plus sirolimus/rapamycin — Study subjects will apply a study product containing polyvinylidene fluoride coating plus 1 mg of sirolimus/rapamycin to either facial angiofibromas or cutaneous neurofibromas
  Arms: NF1 1% Arm; TSC 1% Arm
Drug: Skinercity plus sirolimus/rapamycin — Study subjects will apply a study product containing polyvinylidene fluoride coating plus 5 mg of sirolimus/rapamycin to either facial angiofibromas or cutaneous neurofibromas
  Arms: NF1 5% Arm; TSC 5% Arm

SUMMARY:
This study is a prospective, randomized, double-blind, placebo-controlled evaluation of the safety of a topically applied formulation of rapamycin to cutaneous fibromatous lesions in subjects with Tuberous Sclerosis Complex (TSC) and Neurofibromatosis I (NF1). Subjects will apply either a Polyvinylidene fluoride (PVDF) coating (Skincerity) containing rapamycin or the PVDF coating alone nightly to fibromatous lesions for a duration of six months.

The primary goal of this study is to evaluate the safety of the topical product in patients with TSC and NF1. The secondary goal of this study is to evaluate the effectiveness of the topical product for treatment of cutaneous fibromatous lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to comply with all trial requirements
* Subject is male or female and over 13 years of age
* Subject has a diagnosis of either TSC or NF1 and has visible fibromatous lesions (angiofibromas or neurofibromas)
* Female subjects of child-bearing potential must not be pregnant and must agree to use appropriate contraceptive methods for the duration of the trial

Exclusion Criteria:

* Subject is currently receiving therapy with rapamycin or sirolimus
* Subject is receiving any form of immunosuppression or has previously experienced immune dysfunction
* Subject is currently participating in or has participated within the last 30 days in any clinical trial involving an investigational drug
* Subject has a known hypersensitivity to either the PVDF coating (Skincerity®) or rapamycin
* Subject is a pregnant or nursing female

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rapamycin level | 6 months
Complete blood count | 6 months
Total cholesterol | 6 months
Dermatologic sensitivity at site of application (pain, erythema, edema, pruritis) | 6 months

SECONDARY OUTCOMES:
Reduction in lesion size and appearance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Koenig, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Hope Northrup, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

REFERENCES:
- [Derived] Koenig MK, Hebert AA, Roberson J, Samuels J, Slopis J, Woerner A, Northrup H. Topical rapamycin therapy to alleviate the cutaneous manifestations of tuberous sclerosis complex: a double-blind, randomized, controlled trial to evaluate the safety and efficacy of topically applied rapamycin. Drugs R D. 2012 Sep 1;12(3):121-6. doi: 10.2165/11634580-000000000-00000. PMID 22934754